CLINICAL TRIAL: NCT05865431
Title: Singlet Oxygen Quantification After Skin Exposure to Ultraviolet A (UVA) Light
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1042064
Record Dates: First submitted 2023-04-07; First posted 2023-05-18 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2023-05

CONDITIONS: Sun Damaged Skin
MeSH Terms: interventions — Zinc Oxide; avobenzone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zinc Oxide, Avobenzone, No Product (Experimental): Participants have zinc oxide, avobenzone, and no product applied to 3 different spots on the forearm and singlet oxygen is measured after UV exposure.
  Interventions: Drug: Zinc Oxide and Avobenzone

INTERVENTIONS:
Drug: Zinc Oxide and Avobenzone — Zinc Oxide is applied to one area of the forearm, Avobenzone is applied to another area of the forearm.

SUMMARY:
The objective of this study is quantification of singlet oxygen species in the skin after exposure to Ultraviolet A (UVA) light

DETAILED DESCRIPTION:
Ultraviolet (UV) radiation can lead to skin damage and cancer. Ultraviolet A (UVA) irradiation is 10 to 100 times more abundant in natural sunlight than ultraviolet B (UVB), thus human skin is exposed to more UVA irradiation daily.UVA irradiation is not completely filtered by clothing and it penetrates deeper into the dermis than UVB, potentially causing more damage. It is believed that skin cancer, photo aging, and skin immunomodulation are mediated by the reactive oxygen species (ROS) that are generated in response to UV radiation. Singlet oxygen (1O2) is one type of ROS. The aim of this study is to quantify the level of singlet oxygen generated in the skin after exposure to UVA radiation. Previous studies have used low dose ultraviolet A1(UVA1) irradiation of 20 J/cm2, which mimics exposure to strong sunlight of approximately two hours. This study will use UVA doses equivalent to or less than what humans are exposed to in daily life. Additionally, the aim is to quantify singlet oxygen produced in individuals of various skin types before and after application of sunscreens containing zinc oxide and avobenzone (sun protection factor 30). To our knowledge, there is no method for quantifying singlet oxygen in human skin after exposure to UVA light. This is a novel method that may help the investigators understand further the protective effects of various skin types, as well as sunscreens.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years and older

Exclusion Criteria:

* Those who are currently smoking or have smoked within the past 3 years.
* Aspirin use
* Multivitamins and supplements that contain vitamin E
* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

PRIMARY OUTCOMES:
Amount of singlet oxygen generated by the left forearm skin (2 cm^2) after exposure to UVA radiation dose of 0.33 J/cm2 | 5 minutes at first visit
Amount of singlet oxygen generated by the left forearm skin (2 cm^2) after exposure to UVA radiation dose of 8.25 J/cm2 | 5 minutes at first visit
Amount of singlet oxygen generated by the left forearm skin (2 cm^2) after exposure to UVA radiation dose of 16.5 J/cm2 | 5 minutes at first visit

SECONDARY OUTCOMES:
Difference in singlet oxygen (as measured by singlet oxygen molecule numbers) generated between individuals of different skin Fitzpatrick skin types | Within 24 hours
Difference in singlet oxygen (as measured by thymidine dimer %) generated between individuals of different skin Fitzpatrick skin types | Within 24 hours
Difference in singlet oxygen generation with avobenzone and zinc oxide sunscreens (sun protection factor 30 and 2mg/cm^2 applied for each) vs control (no sunscreen) after exposure to 444.1millijoules (mJ) /cm2 UVA exposure | Within 24 hours
  Difference in singlet oxygen generation (as measured by thymidine dimer %) with two different sunscreens (zinc oxide and avobenzone, each sun protection factor 30 and 2mg/cm^2 applied) vs control (no sunscreen) after exposure to 444.1mJ/cm2 UVA exposure
Difference in singlet oxygen generation with avobenzone and zinc oxide sunscreens (sun protection factor 30 and 2mg/cm^2 applied for each) vs control (no sunscreen) after exposure to 444.1millijoules (mJ) /cm2 UVA exposure | Within 24 hours
  Difference in singlet oxygen generation (as measured by singlet oxygen molecule numbers) with two different sunscreens (zinc oxide and avobenzone, each sun protection factor 30 and 2mg/cm^2 applied) vs control (no sunscreen) after exposure to 444.1mJ/cm2 UVA exposure
Change in appearance of skin pigmentation as measured by colorimetry after UVA exposure | Within 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

REFERENCES:
- [Background] Tewari A, Grage MM, Harrison GI, Sarkany R, Young AR. UVA1 is skin deep: molecular and clinical implications. Photochem Photobiol Sci. 2013 Jan;12(1):95-103. doi: 10.1039/c2pp25323b. PMID 23192740
- [Background] Langstaff SR. Nursing care study. Rheumatoid arthritis treated with penicillamine. Nurs Times. 1975 Jun 12;71(24):918-9. No abstract available. PMID 166356
- [Background] Menter JM, Hatch KL. Clothing as solar radiation protection. Curr Probl Dermatol. 2003;31:50-63. doi: 10.1159/000072237. PMID 12882019
- [Background] Wang F, Smith NR, Tran BA, Kang S, Voorhees JJ, Fisher GJ. Dermal damage promoted by repeated low-level UV-A1 exposure despite tanning response in human skin. JAMA Dermatol. 2014 Apr;150(4):401-6. doi: 10.1001/jamadermatol.2013.8417. PMID 24305962
- [Background] Sklar LR, Almutawa F, Lim HW, Hamzavi I. Effects of ultraviolet radiation, visible light, and infrared radiation on erythema and pigmentation: a review. Photochem Photobiol Sci. 2013 Jan;12(1):54-64. doi: 10.1039/c2pp25152c. PMID 23111621
- [Background] Hanson KM, Clegg RM. Observation and quantification of ultraviolet-induced reactive oxygen species in ex vivo human skin. Photochem Photobiol. 2002 Jul;76(1):57-63. doi: 10.1562/0031-8655(2002)0762.0.co;2. PMID 12126308

DOCUMENTS (1):
  • Study Protocol (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT05865431/Prot_000.pdf